CLINICAL TRIAL: NCT01932567
Title: Effect of Physiotherapy Evaluated by Electrical Impedance Tomography
Brief Title: Electrical Impedance Tomography (EIT) and Physiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, G.Reychler, PhD, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: physioEIT
Record Dates: First submitted 2013-08-19; First posted 2013-08-30 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Respiratory Disease
MeSH Terms: conditions — Respiration Disorders | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Positive expiratory pressure (Experimental): Use of positive expiratory pressure during 3 minutes
  Interventions: Other: Physiotherapy; Procedure: Electrical impedance tomography
- Incentive spirometry (Experimental): Use of incentive spirometry during 3 minutes
  Interventions: Other: Physiotherapy; Procedure: Electrical impedance tomography
- manual airway clearance technique (Experimental): Use of manual airway clearance technique during 3 minutes
  Interventions: Other: Physiotherapy; Procedure: Electrical impedance tomography

INTERVENTIONS:
Other: Physiotherapy
Procedure: Electrical impedance tomography

SUMMARY:
To compare the effect of different airway clearance techniques on lung ventilation by electrical impedance tomography.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Surgery under anesthesia (PEP and incentive spirometry) or healthy subjects
* Intervention time before first bed lift
* Cooperative
* Can perform devices techniques correctly

Exclusion Criteria:

* Patients with pacemaker, implantable pumps or automatic implantable cardioverter defibrillator
* Patients with pulmonary disease (acute or chronic)
* Patients with cognitive problems
* Presence of patches or wounds in EIT belt zone placement
* Patients with initial pain > 2/10
* Patients with severe obesity (BMI > 35)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Regional lung ventilation measured by Electrical impedance tomography | Recording by electrical impedance tomography will be performed during 30 minutes

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Clinique universitaire Saint-Luc, Brussels
  - Cliniques universitaires Saint-Luc, Brussels